CLINICAL TRIAL: NCT05486780
Title: The Effect of Digital Window on Day and Night Perception Status and Sleep Quality in Intensive Care Patients: A Randomized Controlled Trial
Brief Title: The Effect of Digital Window on Day and Night Perception Status and Sleep Quality in Intensive Care Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, ikbal bezek, Master Student, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ilkbal-dw
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Coronary Artery Diseases; Heart Valve Diseases
Keywords: intensive care units; daylight; postoperative patient; sleep quality; clinical trial
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital window (Experimental): The patients who will be assigned to the experimental group will sleep on the 1st, 2nd, and 3rd beds. Experimental group patients are in the field of view of the digital window. A digital window is a tool designed by the researcher to enable patients to differentiate between day and night.
  Interventions: Behavioral: Digital Window
- Control group (No Intervention): the patients who will be assigned to the control group will sleep in the 4th, 5th, and 6th beds. Control group patients are not in the field of view of the digital window. Data collection will be completed by the researcher by completing the Day and Night Perception Form and the Richards Campbell Sleep Scale (Post-Test) on the 1st, 2nd, and 3rd days of post-op for the patients in the control group who are not in the field of view of the digital window.

INTERVENTIONS:
Behavioral: Digital Window — For the digital window, a regal brand, 43R654FC, 43-inch (109 cm) television was used. A three-dimensional frame was built to give the appearance of a window around the television. For the digital window, a regal brand, 43R654FC, 43-inch (109 cm) television was used. A three-dimensional frame was built to give the appearance of a window around the television. Data collection will be completed by the researcher completing the Day and Night Perception Form and the Richards Campbell Sleep Scale (Post-Test) on the 1st, 2nd, and 3rd days of post-op for the patients in the experimental group who are in the field of view of the digital window.
  Arms: Digital window

SUMMARY:
The research will be carried out in the Cardio Vascular Surgery (CVS) Intensive Care Unit (ICU) of Ankara Training and Research Hospital (TRH) . Patients will be divided into two Experimental (n=24) and control (n=24) groups. Simple randomization method will be used in the study, provided that there are equal numbers of male and female patients in the experimental and control groups, regardless of the age of the patients. Patients in the experimental group will use a digital window. The "Patient Information Form","Richard-Campbell Sleep Questionnaire_RCSQ " and " Day and Night Perception Form" will be used in the data collection phase. Ethics committee approval was received from Ankara Yıldırım Beyazıt University Ethics Committee in order to conduct the study.

DETAILED DESCRIPTION:
This research will be carried out as a randomized controlled experimental study to investigate the effect of the digital window on day and night perception status and sleep quality in intensive care patients. The research population consists of patients who underwent CABG and heart valve surgery and were admitted to the CVC ICU of Ankara Training and Research Hospital.

Sample size calculation

In order to calculate the sample size, a pilot study was conducted with 6 patients, three in the experimental group and three in the control group, and these pilot study data were used. As a result of the power analysis made with the help of the G*Power 3.0.10 program, the power of the study was found to be 80% for 2 groups and 3 repetitive study designs with an f=0.20 effect size and 5% margin of error. As a result, at least 42 samples in total, 21 of which were in the experimental group and 21 in the control group, were found to be sufficient. Considering that the sample size obtained is the lowest limit and the patients have the possibility of going into delirium under intensive care conditions or giving up on continuing to work afterward, considering that the losses may be high, 15% of the number determined according to the sampling calculation was calculated and 48 patients who met the criteria for inclusion in the study were sampled. In experimental studies, it is recommended that the sample loss should not be more than 10-15%.

Randomization

A simple randomization method will be used in the study, provided that there are equal numbers of male and female patients in the experimental and control groups, regardless of the age of the patients. Whether the first female and first male patients who will come at the beginning of the study will be in the experimental group or the control group will be determined by drawing lots. The following patients will be divided into two groups, according to the order of arrival, the same-sex patients in the experimental group and the control group.

Data collection tools: The data in the research; Patient Information Form, Richard-Campbell Sleep Questionnaire_RCSQ will be collected using the Day and Night Perception Form.

Research Implementation

Whether the first female and first male patients to come to the CVS ICU on the day of surgery will be the experimental group or the control group will be determined by drawing lots. The following patients will be divided into two groups, according to the order of arrival, same-sex patients in the experimental group and the control group. In this way, it is planned to establish a balance between the groups according to gender. The patients who will be assigned to the experimental group will sleep on the 1st, 2nd, and 3rd beds, and the patients who will be assigned to the control group will sleep in the 4th, 5th, and 6th beds. Data collection will be completed by the researcher by completing the Day and Night Perception Form and the Richards Campbell Sleep Scale (Post-Test) on the 1st, 2nd and 3rd days of post-op for the patients in the experimental group who are in the field of view of the digital window and the patients in the control group who are not in the field of view of the digital window. Night and Day Perception Form will be administered twice a day, once in the morning and in the evening, and Richards Campbell Sleep Scale will be administered once in the morning to each patient at the same time interval.

ELIGIBILITY:
Inclusion Criteria:

* The patient has CABG and heart valve surgery
* The patient's willingness to participate in the study voluntarily
* Patient's ability to answer research questions
* The patient's age range is 19-79
* Being in the post-op period and staying in the ICU for at least 48 hours after the post-op period
* Determined as a Glasgow Coma Scale (GCS) score of 9 or higher

Exclusion Criteria:

* Patient undergoing another operation other than CABG and heart valve surgery
* The patient is intubated
* The patient's use of sedating drugs
* The patient is in delirium
* Patient's age other than 19-79
* Staying in the ICU for less than 48 hours after the post-op period
* Determined as GKS score below 9

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Research shows that gender affects sleep quality in patients with heart valve and coronary artery disease. Therefore, we will randomize participants into the groups, which were similar in terms of gender.
Enrollment: 48 (Estimated)
Dates: Start 2022-08-08 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-01-10 (Estimated)

PRIMARY OUTCOMES:
1.Change in sleep quality | Baseline measurements (Pre-op), at the post-op 1., 2. and 3. days after the completion of the interventions
  Sleep quality will be measured based on the patient report by Richard-Campbell Sleep Questionnaire. A higher score means an increase in sleep quality.
2. Change in day and night perception status | Measurements at the post-op 1., 2. and 3. days after the completion of the interventions
  Day and night perception status will be measured based on the patient report byDay and Night Perception Form.

CONTACTS AND LOCATIONS:
Overall Officials: İlkbal Bezek, Master Student, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Training and Research Hospital-Cardiovascular Surgery Intensive Care Unit, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The confidentiality of the data used in the study will be protected.